CLINICAL TRIAL: NCT06617221
Title: Alveolar Ridge Preservation Using a Composite Graft Plug: Radiographic and Clinical Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Arwa Abubakr Badahdah, Assistant professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC 4350-444
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Extraction Socket Healing; Socket Preservation; Alveolar Ridge Preservation
MeSH Terms: interventions — Transplantation, Homologous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Composite graft plug (Experimental): composite graft plug was placed in the socket after extraction
  Interventions: Biological: Composite graft plug
- Allograft (Active Comparator): allograft was placed in the socket after extraction
  Interventions: Biological: Allograft

INTERVENTIONS:
Biological: Composite graft plug — after tooth extraction the socket was grafted with a composite graft plug
  Arms: Composite graft plug
Biological: Allograft — after tooth extraction the socket was grafted with allograft
  Arms: Allograft

SUMMARY:
The goal of this clinical trial is to determine whether a graft material introduced recently (test) to be used in extraction sockets is as good as a previously known graft material (control) in adults undergoing tooth extraction of a single-rooted tooth.

The main question it aims to answer is:

Is this graft material able to maintain good bone volume and composition after extraction?

Researchers will compare this new graft to a well-studied graft material.

Participants will be randomly assigned to one of the groups and will receive the allocated graft after tooth extraction. The dimension of the alveolar ridge, which supports teeth in the jaw, will be measured before extraction and four months after healing. A cone beam CT Scan will also be obtained.

DETAILED DESCRIPTION:
Alveolar ridge resorption after tooth extraction poses a substantial obstacle for subsequent implant placement, frequently necessitating ridge augmentation treatments. Alveolar ridge preservation (ARP) is intended to reduce these dimensional alterations. Various grafting materials have been used for ARP, with varying success rates in maintaining ridge dimensions. This study compares the clinical and radiological outcomes of a composite graft plug of bioactive resorbable calcium apatite crystals embedded in a collagen matrix to a typical allograft.

This randomized controlled clinical experiment comprised 26 people needing a single-rooted tooth extracted. They were divided into two groups: composite plug and allograft. Clinical measures of soft tissue were collected at baseline and four months after extraction using a stent with reference points. At baseline and four months after extraction, radiographic examinations were performed using cone beam computed tomography (CBCT).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* planned for extraction and alveolar ridge preservation of a single-rooted tooth - -- healthy or have well-controlled systemic disease
* good oral hygiene
* healthy periodontium or at least at the extraction area.

Exclusion Criteria:

* smoking ≥10 cigarettes per day
* generalized periodontitis
* poor oral hygiene
* uncontrolled systemic diseases such as diabetes
* pregnancy
* history of anti-resorptive therapy such as bisphosphonate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
clinical and radiographic ridge alterations | four months
  Using a standardized stent with reference points , the following horizontal clinical measurements were obtained before extraction through the stent holes: buccal soft tissue thickness at 4, 7, and 10 mm apical to the gingival margin and palatal or lingual soft tissue thickness at similar sites. Vertical measurements were obtained an incisal or occlusal hole to the buccal aspect of the ridge (inciso-buccal) and the palatal/ lingual aspect (inciso-palatal). Radiographic width of the alveolar ridge was measure at the same reference points.
  theses measurements were taken at baseline (before extraction) and at 4 months after extraction and socket graft

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz University, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Age, Medical condition, gender
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Jafarian J, Shahrabi-Farahani S, Ferreira CF, Stewart CW, Luepke P. Histological Evaluation of Alveolar Ridge Preservation Using Different Bone Grafts: Clinical Study Analysis Part II. J Oral Implantol. 2024 Jun 1;50(3):260-265. doi: 10.1563/aaid-joi-D-23-00060. PMID 38660739
- [Background] Jones K, Williams C, Yuan T, Digeorge-Foushee AM, Chambers Wilson R, Burton T, Hamlin N, Martinez L. Comparative in vitro study of commercially available products for alveolar ridge preservation. J Periodontol. 2022 Mar;93(3):403-411. doi: 10.1002/JPER.21-0087. Epub 2021 Jul 12. PMID 34114665